CLINICAL TRIAL: NCT03509870
Title: Uncontrolled Non-randomised Single Dose Study of Topically Applied Bone Marrow Derived Allogeneic Mesenchymal Stromal Cells (REDDSTAR (ORBCEL-M)) in Patients With Non-healing Neuroischaemic Diabetic Foot Wounds'
Brief Title: Bone Marrow Derived Allogeneic Mesenchymal Stromal Cells to Non-healing Diabetic Foot Wounds
Acronym: REDDSTAR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study stopped because of lack of recruitment
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-005580-16
Record Dates: First submitted 2018-04-11; First posted 2018-04-26 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetes
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: unblinded single arm intervention
Masking Description: open
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mesenchymal stromal cells (Other): mesenchymal stromal cells in collagen scaffold
  Interventions: Biological: mesenchymal stromal cells

INTERVENTIONS:
Biological: mesenchymal stromal cells — mesenchymal stromal cells in a collagen scaffold

SUMMARY:
examine safety of topical application of single dose allogeneic bone marrow derived mesenchymal stromal cells to non-healing diabetic foot ulcers

DETAILED DESCRIPTION:
1.1 Trial Phase

Phase 1b

1.2 Trial Aims and Objectives

To examine the safety of topical application of a single dose of allogeneic bone marrow derived mesenchymal stromal cells (REDDSTAR ORBCEL-M) seeded in a collagen scaffold to patients with non-healing neuroischaemic diabetic foot wounds.

1.3 Patient Population

Patients with non-healing neuroischaemic diabetic foot wounds despite standard care.

1.4 Trial Setting

Steno Diabetes Center Copenhagen, Denmark and Zelo Phase I Unit, Bispebjerg Hospital, Copenhagen, Denmark.

1.5 Trial Intervention

Topical application of allogeneic bone marrow derived mesenchymal stromal cells seeded in a collagen scaffold to patients with non-healing neuroischaemic diabetic foot wounds.

1.6 Concurrent Control

Open label, uncontrolled, non-randomised, single dose study.

1.7 Sample Size

9

1.8 Method of Participant Assignment

Administration of a single dose of allogeneic bone marrow-derived mesenchymal stromal cells seeded in a collagen scaffold.

1.9 Examination Points

0, 1 week, 2 weeks, 3 weeks, 4 weeks up until 12 weeks or until complete wound closure. After the week 12 visit, or ulcer closure, whichever occurs first, each patient will return to the clinic 1 (± 2 days), 2 (± 2 days), 4 (± 3 days), 8 (±3 days), and 12 (±3days) weeks later for follow-up visits to for adverse events, assess wound, wound closure and durability.

1.10 Primary Outcome

Serious adverse events that are attributable to intervention.

1.11 Secondary Outcomes

Time to complete wound closure (defined as from treatment day 1 to the first visit when closure is documented). Absolute and percent changes in wound area from baseline, at weekly intervals throughout. Durability of wound closure as measured at 4 week intervals for 12 weeks from date of wound closure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Type 1 or Type 2 diabetes mellitus (with any kind or combination of pharmacological treatment for disease and/or complications to disease).
3. HbA1c ≤ 97 mmol/mol (≤ 11%).
4. Males or non-pregnant females.
5. Understand trial information document.
6. Provide written informed consent.
7. Duration of (diabetic foot) wound > 4 but < 52 weeks.
8. Reduction of < 50% area over 4 weeks despite standard care (standard care; off-loading, weekly debridement, dressings, orthotic).
9. Wound area with sharp debridement of ≥ 0.5 but ≤ 4.0 cm2.
10. Clinically non-infected wound.
11. Texas wound stage 1a, 1c or 2a.
12. Location of wound below malleolus.
13. Affected limb toe pressure ≥ 40 mmHg.
14. An ankle-brachial systolic pressure index between 0.7 and 1.3.
15. Diagnosis of peripheral neuropathy using American Diabetes Association guidelines (monofilament/vibration sensation/biothesiometer).
16. Able to adhere to study visit protocol.
17. Adhere to offloading devices/orthotic.

Exclusion Criteria:

1. Life expectancy of less than 12 months.
2. Patients with a definite diagnosis of any immunodeficiency disorder.
3. Viral hepatitis [patient must have negative hepatitis B surface-antigen (HBsAg) and hepatitis C antibody (HepCAb) test results obtained within 2 weeks prior to the Treatment Day (Day 1)].
4. Active, uncontrolled connective tissue disease.
5. Renal failure as defined by serum creatinine > 220 µmol/L.
6. Liver function tests that are > 2.0 times Upper Limit Normal.
7. Poor nutritional status as measured by serum albumin < 30 g/L.
8. Active cancer or a history of cancer in the 5 years prior to signing the informed consent form (history of basal cell carcinoma is allowed).
9. Active wound infection (i.e. recent onset of erythema, oedema, and increased temperature of the foot with normal radiographs).
10. Diabetic Charcot neuroarthropathy or other structural deformity that would prevent adequate off-loading of the study foot.
11. Treatment with any systemic corticosteroid immunosuppressive chemotherapeutic agent, antiviral, or previous/current radiation therapy to lower extremity to be treated within 30 days prior to signing the informed consent form.
12. Having received another investigational drug or biologic within 30 days prior to signing the informed consent form or currently participating in an investigational drug or biologic study.
13. A psychiatric condition or chronic alcohol or drug abuse problem, determined from the patient's medical history, which in the Investigator's opinion may pose a threat to patient compliance.
14. History of non-compliance with treatment or clinical visit attendance (i.e. this study requires that patients will comply with the protocol and ulcer care regimen).
15. Any unstable medical condition judged by the Principal Investigator that would cause the study to be detrimental to the patient.
16. Wounds caused primarily by untreated vascular insufficiency, or where patients are primarily eligible for vascular intervention to promote wound healing.
17. Wounds with an aetiology not related to diabetes.
18. More than three wounds on the target lower extremity.
19. The wound to be studied not anatomically distinct from another wound(s) (separated by < 1 cm from another wound or would interfere with standard of care treatment of another wound. Only one single wound per one study subject can be treated in this study.
20. Wounds which decrease in area by > 50% during the screening 4-week run-in period.
21. Ulcers with underlying osteomyelitis on the leg with the wound to be treated.
22. Patients presenting with the clinical characteristics of cellulitis at the wound site (suppurative inflammation involving particularly the subcutaneous tissue, often mild erythema, tenderness, malaise, chills and fever).
23. Revascularization surgery on the leg with the wound to be treated ≤8 weeks prior to signing the informed consent form.
24. Surgery to lengthen Achilles tendon on the leg with the wound to be treated ≤8 weeks prior to signing the informed consent form.
25. Necrosis, purulence, or sinus tracts that cannot be removed by debridement on foot to be treated.
26. Received dermal substitute or living skin equivalent within 30 days prior to signing the informed consent form.
27. Received prior (Regranex®/becaplermin) therapy within 30 days prior to signing the informed consent form.
28. Has known history of clinical sensitivity reactions to products of bovine origin or to the primary or secondary dressings used in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
serious adverse events attributable to intervention | 24 weeks
  1. Death
  2. Septicaemia
  3. Amputation of the limb administered with therapy
  4. Worsening of the ulcer of the limb administered with therapy
  5. Allergic reaction or anaphylaxis
  6. Abnormal laboratory results
  7. Local or systemic reaction requiring hospital admission

SECONDARY OUTCOMES:
healing | 24 weeks
  time to complete wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided